CLINICAL TRIAL: NCT07360912
Title: Open Haemorrhoidectomy Combined With Lateral Internal Sphincterotomy Versus Conventional Haemorrhoidectomy: A Prospective Randomized Comparative Study
Brief Title: Haemorrhoidectomy With vs Without Lateral Internal Sphincterotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Alaa Alsalaumy, Assistant Professor and Consultant Surgeon, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HLS-RCT-2024
Record Dates: First submitted 2026-01-13; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Grade III and IV Hemorrhoids
Keywords: Hemorrhoids; Hemorrhoidectomy; Lateral Internal Sphincterotomy; Postoperative Pain; Postoperative Bleeding
MeSH Terms: conditions — Lymphoma, Follicular; Hemorrhoids; Pain, Postoperative; Postoperative Hemorrhage | interventions — Hemorrhoidectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hemorrhoidectomy With LIS (Experimental): Patients undergo open hemorrhoidectomy combined with lateral internal sphincterotomy to reduce postoperative pain and anal sphincter spasm.
  Interventions: Procedure: Hemorrhoidectomy With LIS
- Conventional Hemorrhoidectomy (Active Comparator): Patients undergo standard open hemorrhoidectomy without lateral internal sphincterotomy.
  Interventions: Procedure: Conventional Hemorrhoidectomy

INTERVENTIONS:
Procedure: Hemorrhoidectomy With LIS — Open excisional hemorrhoidectomy combined with lateral internal sphincterotomy to reduce anal sphincter spasm and postoperative pain.
  Arms: Hemorrhoidectomy With LIS
Procedure: Conventional Hemorrhoidectomy — Standard open excisional hemorrhoidectomy without lateral internal sphincterotomy.
  Arms: Conventional Hemorrhoidectomy

SUMMARY:
Hemorrhoids are a common anorectal condition that often require surgical treatment in advanced stages. Open hemorrhoidectomy is effective but is frequently associated with significant postoperative pain and early bleeding. Increased anal sphincter spasm after surgery is believed to be a major contributor to these complications.

This study evaluates whether adding lateral internal sphincterotomy (LIS) to conventional open hemorrhoidectomy reduces postoperative pain and bleeding. A total of 120 adult patients with Grade III or IV hemorrhoids were randomized to undergo either open hemorrhoidectomy with LIS or open hemorrhoidectomy alone. Postoperative pain was assessed using a visual analogue scale, and postoperative bleeding was recorded at 24 hours, 48 hours, one week, and two weeks after surgery.

The results of this trial aim to determine whether the addition of LIS provides better short-term recovery and improved postoperative outcomes compared with standard hemorrhoidectomy.

DETAILED DESCRIPTION:
This was a prospective, randomized, comparative clinical trial conducted at Baghdad Teaching Hospital, Iraq, between March 2024 and July 2025. Adult patients aged 18 to 70 years with symptomatic Grade III or IV hemorrhoids were eligible for inclusion. Patients with other anorectal diseases, previous anorectal surgery, inflammatory bowel disease, malignancy, or significant comorbidities were excluded.

A total of 120 patients were randomly assigned into two groups using sealed opaque envelopes. Group A underwent open hemorrhoidectomy combined with lateral internal sphincterotomy, while Group B underwent open hemorrhoidectomy alone. All procedures were performed under general anesthesia by the same experienced surgeon to maintain procedural consistency.

Postoperative pain was assessed using a visual analogue scale at 24 hours, 48 hours, one week, and two weeks after surgery. Postoperative bleeding was recorded at the same time points. Standard postoperative care, including analgesia and sitz baths, was provided to all patients.

The primary outcome was the proportion of patients who were pain-free at one week after surgery. Secondary outcomes included postoperative bleeding at all follow-up time points. The study aimed to evaluate whether the addition of lateral internal sphincterotomy improves early postoperative recovery compared with conventional hemorrhoidectomy alone.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 70 years

  * Patients diagnosed with grade III or IV hemorrhoids
  * Patients scheduled for open hemorrhoidectomy
  * Patients able to provide informed consent

Exclusion Criteria:

* Patients with inflammatory bowel disease
* Patients with anal fissure, fistula, or anorectal malignancy
* Patients with previous anorectal surgery
* Patients with bleeding or coagulation disorders
* Patients unfit for surgery or general or spinal anesthesia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain | Postoperative day 1, day 2, day 7, and day 14
  Pain intensity after hemorrhoidectomy measured using a Visual Analog Scale (VAS, 0-10).

SECONDARY OUTCOMES:
Postoperative bleeding | Postoperative day 1, day 2, day 7, and day 14
  Postoperative bleeding was recorded as the presence or absence of bleeding from the surgical site after hemorrhoidectomy.

CONTACTS AND LOCATIONS:
Overall Officials: Alaa Alsalaumy, Master degree, Principal Investigator — University of baghdad, college of medicine
Locations (1):
- University of baghdad collage of medicine, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the dataset contains confidential clinical information and there is no public data repository for this study.

REFERENCES:
- See also: ClinicalTrials.gov study record — https://clinicaltrials.gov